CLINICAL TRIAL: NCT02705872
Title: Comparison of Two Methods of Administration of the Epidural, by Programmed Intermittent Bolus or Continuous Perfusion, on the Incidence of Cesarean Sections and Instrumented Deliveries in Primiparous Women
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in guidelines
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Philippe VAN DER LINDEN, Head of clinic, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUB-PIB
Record Dates: First submitted 2016-03-02; First posted 2016-03-11 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: First Child Delivery With Epidural
Keywords: Epidural; Programmed intermittent boluses; Cesarian section; Instrumented delivery
MeSH Terms: interventions — Levobupivacaine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Programmed intermittent boluses (Experimental): Epidural analgesia performed with programmed intermittent boluses.
  Interventions: Drug: Chirocaine 0.07% + Sufentanil 0.3 mcg/ml 10ml each 60 minutes
- Continuous perfusion (Active Comparator): Epidural analgesia performed with a continuous perfusion.
  Interventions: Drug: Chirocaine 0.07% + Sufentanil 0.3 mcg/ml 10ml/h

INTERVENTIONS:
Drug: Chirocaine 0.07% + Sufentanil 0.3 mcg/ml 10ml/h — Continuous epidural perfusion: Chirocaine 0.07% + Sufentanil 0.3 mcg/ml with a 10ml/hour rate
  Arms: Continuous perfusion
Drug: Chirocaine 0.07% + Sufentanil 0.3 mcg/ml 10ml each 60 minutes — Injection of programmed intermittent boluses in the epidural space, without continuous perfusion, of the same solution (Chirocaine 0.07% + Sufentanil 0.3 mcg/ml): 10ml each 60 minutes
  Arms: Programmed intermittent boluses

SUMMARY:
The epidural has been recognized for many years as the most effective analgesia method for obstetrical labor. Several different administration protocols have been evaluated over the years with the aim of reducing side effects.

Epidurals have been incriminated in the increase of instrumented births. It is indeed possible that the motor block induced by the epidural reduces the pelvic tonus and the ability of the mother to push during the second stage of the labor. Furthermore, this motor block might lead to a ill rotation of the foetal head within the pelvis, which could lead to instrumentation (suction cups, forceps).

In the investigator's institution, an ongoing study also provided interim that showed that the use of a low concentration of local anesthetics (as opposed to a higher concentration) tends to decrease the instrumentation and cesarean sections rate in the institution's population.However, the optimal administration mode of the local anesthetic in the epidural remains unknown.

In the last few years, there has been a growing interest for a new method of administration of the solution within the epidural, by programmed intermittent bolus. This method allows a better distribution of the local anesthetics in the epidural space, compared to a continuous perfusion.

This study therefore focuses on the relationship between the use of epidural with programmed intermittent boluses and the rate of instrumented deliveries and cesarean sections.

The exact mode of administration of boluses is also subject to discussion in the literature. One can question whether it is preferable to administer smaller boluses more frequently or larger less frequent boluses. A few studies have investigated this issue and recommend to administer larger and more spaced bolus (10 mL to 60 minutes).This better matches the sought after physiology (ie a wider distribution in the epidural space) and provides equivalent analgesia to smaller, more frequent boluses.

DETAILED DESCRIPTION:
The epidural has been recognized for many years as the most effective analgesia method for obstetrical labor. Several different administration protocols have been evaluated over the years with the aim of reducing side effects.

Epidurals have been incriminated in the increase of instrumented births. It is indeed possible that the motor block induced by the epidural reduces the pelvic tonus and the ability of the mother to push during the second stage of the labor. Furthermore, this motor block might lead to a ill rotation of the foetal head within the pelvis, which could lead to instrumentation (suction cups, forceps).

In 2001, the COMET study showed that the use of low anesthetics concentrations decreases the motor bloc and allows to increase the rate of vaginal deliveries and decrease the rate of instrumented births.

In the investigator's institution, an ongoing study also provided interim that showed that the use of a low concentration of local anesthetics (as opposed to a higher concentration) tends to decrease the instrumentation and cesarean sections rate in the institution's population.

However, the optimal administration mode of the local anesthetic in the epidural remains unknown.

In the last few years, there has been a growing interest for a new method of administration of the solution within the epidural, by programmed intermittent bolus. This method allows a better distribution of the local anesthetics in the epidural space, compared to a continuous perfusion.

Several studies have been performed and show that this mode of administration allows to decrease the local anesthetics injected dosis and gives a better maternal satisfaction. A meta-analysis performed in 2013 also shows a tendency towards the decrease of instrumented deliveries with this method. Sadly, no studies up to this date have the needed power to prove this point with certainty.

This study therefore focuses on the relationship between the use of epidural with programmed intermittent boluses and the rate of instrumented deliveries and cesarean sections.

The exact mode of administration of boluses is also subject to discussion in the literature. One can question whether it is preferable to administer smaller boluses more frequently or larger less frequent boluses. A few studies have investigated this issue and recommend to administer larger and more spaced bolus (10 mL to 60 minutes).This better matches the sought after physiology (ie a wider distribution in the epidural space) and provides equivalent analgesia to smaller, more frequent boluses.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age
* Primiparous
* Pregnancy over 36 weeks of gestational age and <42 weeks of gestational age
* Written informed consent
* Cervical dilatation between 3 and 6 cm at recruitment
* Single pregnancy
* Foetus in cephalic position

Exclusion Criteria:

* Participation refusal or epidural contra-indication
* Multiparous
* Allergy to the products used
* Twin pregnancy
* Height <1m55 and/or narrow pelvis, as shown by imagery
* Language barrier
* Patients with a BMI superior or equal to 35 (computed with the weight at the beginning of the pregnancy)
* Cervical dilatation at recruitment <3 or >6 cm
* ASA score (American Society of Anesthesiologists) 3 or 4
* Foetus in transverse or seat position

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Rate of instrumented deliveries (suction pumps, forceps) | 24h after the baby's birth
  Number of deliveries requiring instrumentation (suction pumps, forceps)
Rate of cesarian sections | 24h after the baby's birth
  Number of deliveries requiring a cesarian section

SECONDARY OUTCOMES:
Number of anesthesist interventions | Starting from the first injection of the epidural till the baby's birth
  Number of visits of the anesthesist, either requested by the patient (request for additional analgesia by the patient because of pain during labor: the pain itself is not measured), either necessary because of side effects (nausea, pruritus).
Maternal satisfaction | 24h after the baby's birth
  Will be assessed by means of a questionnaire (0 to 100 visual scale)
Presence of a motor block | At the precise moment when the cervix reaches complete dilatation (10 cm opening) during labor
  Assessed by the anesthesist with the Bromage modified scale

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] Howell CJ. Epidural versus non-epidural analgesia for pain relief in labour. Cochrane Database Syst Rev. 2000;(2):CD000331. doi: 10.1002/14651858.CD000331. PMID 10796196
- [Background] George RB, Allen TK, Habib AS. Intermittent epidural bolus compared with continuous epidural infusions for labor analgesia: a systematic review and meta-analysis. Anesth Analg. 2013 Jan;116(1):133-44. doi: 10.1213/ANE.0b013e3182713b26. Epub 2012 Dec 7. PMID 23223119
- [Background] Thorp JA, Hu DH, Albin RM, McNitt J, Meyer BA, Cohen GR, Yeast JD. The effect of intrapartum epidural analgesia on nulliparous labor: a randomized, controlled, prospective trial. Am J Obstet Gynecol. 1993 Oct;169(4):851-8. doi: 10.1016/0002-9378(93)90015-b. PMID 8238138
- [Background] Comparative Obstetric Mobile Epidural Trial (COMET) Study Group UK. Effect of low-dose mobile versus traditional epidural techniques on mode of delivery: a randomised controlled trial. Lancet. 2001 Jul 7;358(9275):19-23. doi: 10.1016/S0140-6736(00)05251-X. PMID 11454372
- [Background] Kaynar AM, Shankar KB. Epidural infusion: continuous or bolus? Anesth Analg. 1999 Aug;89(2):534. doi: 10.1097/00000539-199908000-00063. No abstract available. PMID 10439786
- [Background] Wong CA, Ratliff JT, Sullivan JT, Scavone BM, Toledo P, McCarthy RJ. A randomized comparison of programmed intermittent epidural bolus with continuous epidural infusion for labor analgesia. Anesth Analg. 2006 Mar;102(3):904-9. doi: 10.1213/01.ane.0000197778.57615.1a. PMID 16492849
- [Background] Sia AT, Leo S, Ocampo CE. A randomised comparison of variable-frequency automated mandatory boluses with a basal infusion for patient-controlled epidural analgesia during labour and delivery. Anaesthesia. 2013 Mar;68(3):267-75. doi: 10.1111/anae.12093. Epub 2012 Dec 20. PMID 23278328
- [Background] Lim Y, Chakravarty S, Ocampo CE, Sia AT. Comparison of automated intermittent low volume bolus with continuous infusion for labour epidural analgesia. Anaesth Intensive Care. 2010 Sep;38(5):894-9. doi: 10.1177/0310057X1003800514. PMID 20865875
- [Background] Wong CA, McCarthy RJ, Hewlett B. The effect of manipulation of the programmed intermittent bolus time interval and injection volume on total drug use for labor epidural analgesia: a randomized controlled trial. Anesth Analg. 2011 Apr;112(4):904-11. doi: 10.1213/ANE.0b013e31820e7c2f. PMID 21430035
- [Background] Breen TW, Shapiro T, Glass B, Foster-Payne D, Oriol NE. Epidural anesthesia for labor in an ambulatory patient. Anesth Analg. 1993 Nov;77(5):919-24. doi: 10.1213/00000539-199311000-00008. PMID 8214727